CLINICAL TRIAL: NCT05845333
Title: Neurocognitive Abnormalities in Stimulant Abuse Among High-Risk Women
Status: Recruiting | Type: Observational
Sponsor: The Mind Research Network (Other)
Responsible Party: Principal Investigator, Kent Kiehl, Professor of Psychology, Neuroscience and Law, Executive Science Officer, The Mind Research Network
Other Study IDs: 15050
Record Dates: First submitted 2023-04-07; First posted 2023-05-06 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Stimulant Abuse; Criminal Behavior
MeSH Terms: conditions — Criminal Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Stimulant Use Severity High
  Interventions: Other: Decision task
- Stimulant Use Severity Medium
  Interventions: Other: Decision task
- Stimulant Use Severity Low
  Interventions: Other: Decision task
- Psychopathic Traits High
  Interventions: Other: Decision task
- Psychopathic Traits Medium
  Interventions: Other: Decision task
- Psychopathic Traits Low
  Interventions: Other: Decision task
- Community (Healthy) Controls
  Interventions: Other: Decision task

INTERVENTIONS:
Other: Decision task — Participants will complete a simple and/or moral decision making functional MRI task.

SUMMARY:
Substance use disorders and psychopathy are serious and costly mental health issues. Psychopathy is known to be associated with aberrant moral decision making and there is considerable interest in determining whether substance use disorders lead to impairments in these same cognitive processes. Recent large-scale research initiatives in forensic settings have begun to identify substance abuse and psychopathy-related disruption in the neural mechanisms involved in moral decision-making processes, and associations between these neural networks and future relapse and antisocial behavior. Here the investigators extend prior work (with incarcerated men) to examine these issues among incarcerated women in order to better understand sex differences. This project addresses the overall lack of neurocognitive research in criminal offenders with substance use disorders, thereby focusing on a major public health issue in an underserved and understudied population.

DETAILED DESCRIPTION:
There continues to be great interest and public health relevance with regard to understanding the neurobiological systems that underlie the comorbidity of substance use disorders and other psychiatric conditions. In a previous award, efforts were focused upon characterizing the neural circuitry underlying moral decision making in incarcerated men with varying levels of two frequently co-occurring conditions: stimulant abuse and psychopathy. Here this work will be extended to incarcerated women, to examine longitudinal outcomes and apply state-of-the-art network analyses for predictive models. Prior studies have demonstrated sex differences in the degree and expression of psychopathic traits, patterns of stimulant abuse, and moral decision-making. However, the neural circuitry that underlies these sex differences is not well understood. Substantial sex differences in regional gray matter volume and density in extant samples have also been identified. Collectively, sex differences in pathophysiology could have significant implications for treatment strategies and differential biomarkers of treatment prediction and outcome in men and women. The investigators will implement the research strategy with a large incarcerated population by deploying a unique mobile MRI scanner to the regional women's prison. Participants will be stratified by level of lifetime stimulant (cocaine, amphetamine) use severity and psychopathic traits (high, medium, low) and will undergo anatomical and functional MRI scanning while completing multi-modal (i.e., linguistic and picture) decision-making tasks. Results will be compared to those obtained in a prior award (incarcerated men, n>300). Functional network and dynamic network connectivity will also be examined in women using a new multiband echo planar imaging (EPI) pulse sequence, and longitudinal outcomes after release to the community will be collected to test behavioral and neuropredictive models of relapse and future antisocial behavior. This work is expected to generate a large, robust dataset that characterizes the overlapping and unique aspects of neural circuitry underlying stimulant use and psychopathy in females and males. The proposed research is in line with recent priorities emphasized by the National Institute on Drug Abuse (NIDA) for projects aimed at examining male-female differences, and effects specific to females, to improve understanding of the nature and etiology of drug abuse.

ELIGIBILITY:
Inclusion Criteria:

* Biological sex is female
* Intelligence Quotient 70 or higher
* Reading level 5th grade or higher
* Able to speak and understand English

Exclusion Criteria:

* Uncorrectable auditory or visual deficits
* Currently pregnant
* MRI contraindication
* Central nervous system disease
* Current major medical condition
* Hypertension with complications (e.g., stroke)
* Diabetes with complications
* Lifetime history of psychotic disorder
* Self-report of psychotic disorder (with psychiatric hospitalization) in first degree relative
* Drug use in past three months

(Healthy controls only):

* History of arrest
* Substance use beyond light alcohol or marijuana use
* Currently taking psychotropic medications

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Incarcerated and non-incarcerated adult women
Sampling Method: Probability Sample
Enrollment: 334 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Gray matter volume during MRI scan & stimulant use | During MRI procedure
  Gray matter volume (using relevant MRI analysis platforms - Statistical Parametric Mapping/SPM) correlation with stimulant use (assessed using a modified version of the Addiction Severity Index)
White matter integrity during MRI scan & stimulant use | During MRI procedure
  White matter integrity (using relevant MRI analysis platforms - Functional Magnetic Resonance Imaging of the Brain software library (FSL)) correlation with stimulant use (assessed using a modified version of the Addiction Severity Index)
Functional brain response during MRI scan & stimulant use during simple linguistic decision task | During MRI procedure
  Functional brain responses (Blood Oxygen Level Dependent/BOLD) (using relevant MRI analysis platforms - SPM, Group Independent Components Analysis Functional Toolbox/GIFT) during Simple Linguistic Decision Task correlation with stimulant use (assessed using a modified version of the Addiction Severity Index)
Functional brain response during MRI scan & stimulant use during simple picture decision task | During MRI procedure
  Functional brain responses (Blood Oxygen Level Dependent/BOLD) (using relevant MRI analysis platforms - SPM, Group Independent Components Analysis Functional Toolbox/GIFT) during Simple Picture Decision Task correlation with stimulant use (assessed using a modified version of the Addiction Severity Index)
Functional brain response during MRI scan & stimulant use during moral linguistic decision task | During MRI procedure
  Functional brain responses (Blood Oxygen Level Dependent/BOLD) (using relevant MRI analysis platforms - SPM, Group Independent Components Analysis Functional Toolbox/GIFT) during Moral Linguistic Decision Task correlation with stimulant use (assessed using a modified version of the Addiction Severity Index)
Functional brain response during MRI scan & stimulant use during moral picture decision task | During MRI procedure
  Functional brain responses (Blood Oxygen Level Dependent/BOLD) (using relevant MRI analysis platforms - SPM, Group Independent Components Analysis Functional Toolbox/GIFT) during Moral Picture Decision Task correlation with stimulant use (assessed using a modified version of the Addiction Severity Index)
Functional connectivity during MRI scan & stimulant use during simple linguistic decision task | During MRI procedure
  Functional connectivity (using relevant analysis MRI platforms - GIFT) during Simple Linguistic Decision Task correlation with stimulant use (assessed using a modified version of the Addiction Severity Index)
Functional connectivity during MRI scan & stimulant use during simple picture decision task | During MRI procedure
  Functional connectivity (using relevant analysis MRI platforms - GIFT) during Simple Linguistic Decision Task correlation with stimulant use (assessed using a modified version of the Addiction Severity Index)
Functional connectivity during MRI scan & stimulant use during moral linguistic decision task | During MRI procedure
  Functional connectivity (using relevant analysis MRI platforms - GIFT) during Moral Linguistic Decision Task correlation with stimulant use (assessed using a modified version of the Addiction Severity Index)
Functional connectivity during MRI scan & stimulant use during moral picture decision task | During MRI procedure
  Functional connectivity (using relevant analysis MRI platforms - GIFT) during Moral Picture Decision Task correlation with stimulant use (assessed using a modified version of the Addiction Severity Index)
Gray matter volume during MRI scan & psychopathic traits | During MRI procedure
  Gray matter volume (using relevant MRI analysis platforms - Statistical Parametric Mapping/SPM) correlation with psychopathic traits (assessed using the Psychopathy Checklist-Revised)
White matter integrity during MRI scan & psychopathic traits | During MRI procedure
  White matter integrity (using relevant MRI analysis platforms - Functional Magnetic Resonance Imaging of the Brain software library (FSL)) correlation with psychopathic traits (assessed using the Psychopathy Checklist-Revised)
Functional brain response during MRI scan & psychopathic traits during simple linguistic decision task | During MRI procedure
  Functional brain responses (Blood Oxygen Level Dependent/BOLD) (using relevant MRI analysis platforms - SPM, Group Independent Components Analysis Functional Toolbox/GIFT) during Simple Linguistic Decision Task correlation with psychopathic traits (assessed using the Psychopathy Checklist-Revised)
Functional brain response during MRI scan & psychopathic traits during simple picture decision task | During MRI procedure
  Functional brain responses (Blood Oxygen Level Dependent/BOLD) (using relevant MRI analysis platforms - SPM, Group Independent Components Analysis Functional Toolbox/GIFT) during Simple Picture Decision Task correlation with psychopathic traits (assessed using the Psychopathy Checklist-Revised)
Functional brain response during MRI scan & psychopathic traits during moral linguistic decision task | During MRI procedure
  Functional brain responses (Blood Oxygen Level Dependent/BOLD) (using relevant MRI analysis platforms - SPM, Group Independent Components Analysis Functional Toolbox/GIFT) during Moral Linguistic Decision Task correlation with psychopathic traits (assessed using the Psychopathy Checklist-Revised)
Functional brain response during MRI scan & psychopathic traits during moral picture decision task | During MRI procedure
  Functional brain responses (Blood Oxygen Level Dependent/BOLD) (using relevant MRI analysis platforms - SPM, Group Independent Components Analysis Functional Toolbox/GIFT) during Moral Picture Decision Task correlation with psychopathic traits (assessed using the Psychopathy Checklist-Revised)
Functional connectivity during MRI scan & psychopathic traits during simple linguistic decision task | During MRI procedure
  Functional connectivity (using relevant analysis MRI platforms - GIFT) during Simple Linguistic Decision Task correlation with psychopathic traits (assessed using the Psychopathy Checklist-Revised)
Functional connectivity during MRI scan & psychopathic traits during simple picture decision task | During MRI procedure
  Functional connectivity (using relevant analysis MRI platforms - GIFT)) during Simple Picture Decision Task correlation with psychopathic traits (assessed using the Psychopathy Checklist-Revised)
Functional connectivity during MRI scan & psychopathic traits during moral linguistic decision task | During MRI procedure
  Functional connectivity (using relevant analysis MRI platforms - GIFT) during Moral Linguistic Decision Task correlation with psychopathic traits (assessed using the Psychopathy Checklist-Revised)
Functional connectivity during MRI scan & psychopathic traits during moral picture decision task | During MRI procedure
  Functional connectivity (using relevant analysis MRI platforms - GIFT) during Moral Picture Decision Task correlation with psychopathic traits (assessed using the Psychopathy Checklist-Revised)
Relapse to/change in stimulant use post-release | Every 3 months post release for duration of grant (5 years)
  Return to stimulant use (assessed using timeline follow back calendar (TLFB)) post-release from incarceration
Return to/change in antisocial behavior post-release | Every 3 months post release for duration of grant (5 years)
  Return to antisocial behavior (assessed via self report and/or official records) post-release from incarceration

CONTACTS AND LOCATIONS:
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States